CLINICAL TRIAL: NCT06945419
Title: A Single-Dose and Multiple-Ascending Dose Study of LY4086940 in Healthy Participants and Participants With Overweight or Obesity, With or Without Type 2 Diabetes
Brief Title: A Study of LY4086940 in Healthy Participants and Participants With Overweight or Obesity, With or Without Type 2 Diabetes
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 27267; J5U-MC-YGAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-04-18; First posted 2025-04-25 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Healthy; Overweight; Obesity; Type 2 Diabetes
Keywords: Oral; Incretin; Weight loss; Overweight; Obesity; Diabetes
MeSH Terms: conditions — Overweight; Obesity; Diabetes Mellitus, Type 2; Weight Loss; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Part A: LY4086940 Single Dose (Healthy Participants) (Experimental): Participants will receive a single dose of LY4086940 orally
  Interventions: Drug: LY4086940
- Part A: Placebo Single Dose (Healthy Participants) (Placebo Comparator): Participants will receive a single dose of placebo orally
  Interventions: Drug: Placebo
- Part A: LY4086940 Multiple Dose (Healthy Participants) (Experimental): Participants will receive LY4086940 orally for 3 days
  Interventions: Drug: LY4086940
- Part A: Placebo Multiple Dose (Healthy Participants) (Placebo Comparator): Participants will receive placebo orally for 3 days
  Interventions: Drug: Placebo
- Part B: LY4086940 Multiple Dose (Participants with Overweight or Obesity) (Experimental): Participants will receive LY4086940 orally for 4 weeks
  Interventions: Drug: LY4086940
- Part B: Placebo Multiple Dose (Participants with Overweight or Obesity) (Placebo Comparator): Participants will receive placebo orally for 4 weeks
  Interventions: Drug: Placebo
- Part C: LY4086940 Multiple Dose (Japanese/Chinese Participants with Overweight or Obesity) (Experimental): Participants will receive LY4086940 orally for 4 weeks
  Interventions: Drug: LY4086940
- Part C: Placebo Multiple Dose (Japanese/Chinese Participants with Overweight or Obesity (Placebo Comparator): Participants will receive placebo orally for 4 weeks
  Interventions: Drug: Placebo
- Part D: LY4086940 Multiple Dose (Participants with Type 2 Diabetes with Overweight or Obesity) (Experimental): Participants will receive LY4086940 orally for 4 weeks
  Interventions: Drug: LY4086940
- Part D: Placebo Multiple Dose (Participants with Type 2 Diabetes with Overweight or Obesity) (Placebo Comparator): Participants will receive placebo orally for 4 weeks
  Interventions: Drug: Placebo
- Part E (Open-Label): LY4086940 Single Dose (Healthy Participants) (Experimental): Participants will receive a single dose of LY4086940 intravenously (IV)
  Interventions: Drug: LY4086940

INTERVENTIONS:
Drug: LY4086940 — Administered orally
  Arms: Part A: LY4086940 Multiple Dose (Healthy Participants); Part A: LY4086940 Single Dose (Healthy Participants); Part B: LY4086940 Multiple Dose (Participants with Overweight or Obesity); Part C: LY4086940 Multiple Dose (Japanese/Chinese Participants with Overweight or Obesity); Part D: LY4086940 Multiple Dose (Participants with Type 2 Diabetes with Overweight or Obesity)
Drug: Placebo — Administered orally
  Arms: Part A: Placebo Multiple Dose (Healthy Participants); Part A: Placebo Single Dose (Healthy Participants); Part B: Placebo Multiple Dose (Participants with Overweight or Obesity); Part C: Placebo Multiple Dose (Japanese/Chinese Participants with Overweight or Obesity; Part D: Placebo Multiple Dose (Participants with Type 2 Diabetes with Overweight or Obesity)
Drug: LY4086940 — Administered IV
  Arms: Part E (Open-Label): LY4086940 Single Dose (Healthy Participants)

SUMMARY:
The main purpose of this study is to evaluate the safety, tolerability of LY4086940 and how it is processed in the body.

Participation in Part A of the study will last about 10 weeks and may include up to 6 visits. Participation in Parts B, C, D will last approximately 15 weeks and may include up to 9 visits. Participation in Part E will last approximately 7 weeks and may include up to 12 visits.

ELIGIBILITY:
Inclusion Criteria:

* Have no significant body weight change for the 3 months prior to screening

Part A and Part E:

* Are considered healthy
* Have a body mass index (BMI) of 22 to 35 kilograms per square meter (kg/m2) at screening

Part B:

* Have a BMI of 27 to 45 kg/m2 at screening

Part C:

* Have a BMI of 25 to 45 kg/m2 at screening

Part D:

* Have type 2 diabetes
* Have hemoglobin A1C (HbA1c) ≥7.0% and ≤10.5% at screening
* Have a BMI of 27 to 45 kg/m2 at screening

Exclusion Criteria:

* Have had an acute cardiovascular condition within the past 6 months prior to screening
* Have liver disease or pancreatitis
* Have used medications for weight loss within the 3 months prior to screening

Parts A, B, C, E:

* Have any form of diabetes

Part D:

* Have type 1 diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 201 (Estimated)
Dates: Start 2025-04-23 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Events (SAE) Considered by the Investigator to be Related to Study Drug Administration | Baseline through Week 15

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of LY4086940 | Predose up to Day 63
PK: Area Under the Concentration Versus Time Curve (AUC) of LY4086940 | Predose up to Day 63

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- United States (3):
  - Fortrea Clinical Research Unit, Daytona Beach, Florida
  - Fortrea Clinical Research Unit, Dallas, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
- Lilly Centre for Clinical Pharmacology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of LY4086940 in Healthy Participants and Participants With Overweight or Obesity, With or Without Type 2 Diabetes — https://trials.lilly.com/en-US/trial/599675